CLINICAL TRIAL: NCT04647357
Title: A Trial of SHR-1316 Maintenance Therapy for Limited Stage Small Cell Lung Cancer Without Progression After First Line Concurrent Chemoradiotherapy Treatment
Brief Title: A Trial of SHR-1316 Maintenance Therapy for Limited Stage Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xiaorong Dong, Director, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LS-SCLC-MT-IIT-SHR1316
Record Dates: First submitted 2020-11-27; First posted 2020-11-30 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Limited-stage Small Cell Lung Cancer, LS-SCLC
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1316 (Experimental)
  Interventions: Drug: SHR-1316

INTERVENTIONS:
Drug: SHR-1316 — Anti-PD-L1 antibody，Maintenance therapy, The drug was administered every three weeks

SUMMARY:
SHR-1316 as Maintenance therapy for limited stage small cell lung cancer without progression after first line platinum based concurrent chemoradiotherapy

ELIGIBILITY:
Inclusion Criteria:

1. The age is 18-75 years old (including both ends), regardless of gender;
2. Histologically confirmed limited stage small cell lung cancer ;
3. ECOG PS 0 ~ 1;
4. Patients received at least 2 cycles of platinum based chemotherapy and radiotherapy, and completed within 1 to 42 days before the first medication.
5. The last chemotherapy must be finished before or at the same time of radiotherapy.
6. The disease did not progress after concurrent chemoradiotherapy;
7. The expected survival time was more than 3 months;
8. Pulmonary function: FEV1 > 70%;

Exclusion Criteria:

1. The subjects volunteered to participate in the study, signed the informed consent form, had good compliance and cooperated with the follow-up.
2. Mixed SCLC or NSCLC confirmed by histology;
3. Locally advanced small cell lung cancer receiving sequential chemoradiotherapy;
4. Have received anti-tumor therapy of systemic immune checkpoint inhibitors for SCLC;
5. Extensive SCLC;
6. Operable SCLC (clinical stage T1-2N0, except for those who are contraindicated or refuse surgery);
7. Interstitial pneumonia
8. History of active, known or suspected autoimmune diseases and autoimmune diseases, including but not limited to myasthenia gravis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc.
9. HIV, active Hepatitis B or Hepatitis C infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-11-27 (Estimated); Primary Completion 2023-05-27 (Estimated); Study Completion 2023-12-27 (Estimated)

PRIMARY OUTCOMES:
PFS | Up to approximately 24 months
  progression-free survival